CLINICAL TRIAL: NCT05164562
Title: Prevalence of Musculoskeletal Disorders of Upper Limb in Type 1 Diabetes Patients
Acronym: TMS-DT1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-013-TMS-DT1
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes
Keywords: musculoskeletal disorders; prevalence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Musculoskeletal Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- type 1 diabetes: "type 1 diabetes" group: patients with type 1 diabetes
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Description: musculoskeletal disorders of upper limb evaluation

SUMMARY:
Osteopenia and osteoporosis, particularly related to insulinopenia, are common in type 1 diabetes and increase the risk of fractures. Musculoskeletal disorders of the upper limb are a common complication of type 1 diabetes. However, there is no official recommendation for screening for musculoskeletal disorders in France.

DETAILED DESCRIPTION:
The aim of the study is to describe prevalence of musculoskeletal disorders of upper limb in type 1 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged of 18 and more
* with type 1 diabetes
* agreeing to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
musculoskeletal disorders of upper limb | Day 0
  musculoskeletal disorders of upper limb evaluated using Quick Dash (Quick Disabilities of Arm, Shoulder and Hand).
  Quick Dash is a 11 items questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level. The score ranges from 0 (no disability) to 100 (most severe disability), a higher score indicates a greater level of disability and severity, whereas, lower score indicates a lower level of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Reims, Reims, Grand Est, France

IPD SHARING:
Plan to Share IPD: No